CLINICAL TRIAL: NCT03553134
Title: Descriptive Study of Brain Velocity in Transcranial Doppler in Newborns Over 35 Weeks of Gestational Age in the Maternity Ward
Acronym: VELOCITE
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: LITZLER-RENAULT 2018 VELOCITE
Record Dates: First submitted 2018-05-29; First posted 2018-06-12 (Actual); Last update posted 2019-09-04 (Actual); Status verified 2019-09

CONDITIONS: Newborn

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: transcranial doppler ultrasound scan — Carried out at 4 different times: at birth, 6, 24 and 48 hours of life (duration: 10 minutes)
Diagnostic Test: ultrasound scan centered on the arterial canal — Carried out at 4 different times: at birth, 6, 24 and 48 hours of life (duration: 5 minutes)

SUMMARY:
There are significant variations in blood circulation at birth with the transition from fetal to permanent circulation. These variations are particularly impacted by the closure of the arterial canal within the first 48 hours of life.

Blood circulation velocity values within the cerebral arteries have been well documented in newborns and infants a few days old. However, the initial values of these velocities and their variations during the first hours of life are not well known.

The objective of this study is to describe the evolution of brain circulation at birth in newborns over 35 weeks of gestational age and to investigate the effect of arterial canal closure on brain circulation.

ELIGIBILITY:
Inclusion Criteria:

* Written consent of parent
* Newborns over 35 weeks of amenorrhoea hospitalized in the maternity ward

Exclusion Criteria:

* person not affiliated to a health insurance scheme
* Sepsis
* Ductal dependent heart disease
* Neurological impairment (anoxoischemic encephalopathy Sarnat>1, pH<7 and/or lactates>11, meningitis)
* Obstetrical trauma (instrumental delivery by forceps, vacuum cup or spatulas)
* Potentially lethal malformation
* Anemia (hemoglobin<14g/dl)
* Polyglobulia (hemoglobin>22g/dl)
* Small for gestational age (weight<10th percentile)
* Large for gestational age (weight>97th percentile)
* Proven gestational diabetes (non-insulin-dependent and insulin-dependent)
* Maternal medical treatment (cardiac or anti-epileptic)
* Inadequate parent understanding

Max Age: 6 Hours | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Newborns over 35 weeks of amenorrhoea
Sampling Method: Non-Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2018-04-19 (Actual); Primary Completion 2018-10-25 (Actual); Study Completion 2018-10-25 (Actual)

PRIMARY OUTCOMES:
Right and left average velocity of the cerebral artery | Change from birth to 48 hours of life

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Dijon Bourogne, Dijon, France